CLINICAL TRIAL: NCT04554134
Title: The First Affiliated Hospital of Nanjing Medical University
Brief Title: The Hybrid Combination of CCTA and SPECT and CAG for Evaluation Prognosis of CAD: an Observational Follow-up Study
Acronym: HSCA
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Huai'an First People's Hospital (Other); Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Xu Zhihui, Director, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2019-SR-242; BK20141020 (Other Grant/Funding Number: Zhihui Xu)
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Coronary Disease
Keywords: SPECT; CCTA; CAG; Hybrid
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 550 patients with stable angina (40-70% stenosis) tested by coronary CT angiography (CCTA) and single photon emission computed tomography (SPECT) and coronary angiography (CAG) within 3 months were retrospectively recruited from 2005 to 2015 and follow up to 5 years. A new hybrid software was used to analysis the image data.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70
2. Gender: All
3. coronary artery disease patients (CAD)
4. underwent CCTA, SPECT and coronary angiography (CAG) together within 3 months
5. Time: 2005-2015

Exclusion Criteria:

1. dilated cardiomyopathy (DCM), hypertrophic cardiomyopathy (HCM), congenital heart disease (CHD), atrial fibrillation (AF), ventricular tachycardia (VT)
2. Prior coronary revascularization;
3. permanent pacemaker or internal defibrillator
4. prosthetic heart valve
5. coronary image lose
6. coronary artery severe calcification
7. motion artifacts and poor CCTA image quality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were suspected coronary artery disease and underwent CCTA, SPECT and CAG within 3 months from 2005 to 2015.
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 5 YEARS
  All-cause death, cardiac death, ischemic stroke, unplanned revascularization and nonfatal myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chai, MD, Study Chair — The First Affiliated Hospital Hospital of Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
The hybrid software will be uploaded to the open internet. Cardiologist could upload their patients' image data and the hybrid results will be proved.